CLINICAL TRIAL: NCT00326105
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group, Placebo- Controlled Phase III Study of the Efficacy and Safety of Quetiapine Fumarate Sustained Release (Seroquel SRTM) in Combination With an Antidepressant in the Treatment of Patients With Major Depressive Disorder With Inadequate Response to an Antidepressant Treatment (PEARL STUDY)
Brief Title: Efficacy and Safety of Quetiapine Fumarate Sustained Release (SEROQUEL SR) in Combination With an Antidepressant in the Treatment of Major Depressive Disorders
Acronym: PEARL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1448C00006; PEARL
Record Dates: First submitted 2006-05-15; First posted 2006-05-16 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Major Depressive Disorder
Keywords: MDD; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine fumarate

SUMMARY:
The purpose of this study is to evaluate the efficacy of quetiapine SR in combination with an antidepressant versus an antidepressant alone in patients with MDD with inadequate response to an antidepressant treatment.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to provide written informed consent before beginning any study related procedures
* Patient has a documented clinical diagnosis of major depressive disorder
* Patient is able to understand and comply with the requirements of the study, as judged by a study investigator

Exclusion Criteria:

* Patients with a history of non-compliance as judged by the study investigator
* Patients with a known lack of response to previous treatment with quetiapine
* Patients who have participated in a clinical trial within 4 weeks of randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2006-04; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of quetiapine SR in combination with an antidepressant versus an antidepressant alone in MDD patients with inadequate response to an antidepressant treatment as assessed by the change from randomization to week 6 in the MADRS

SECONDARY OUTCOMES:
To evaluate if quetiapine SR in combination with an antidepressant improves health-related quality of life of patients with MDD, compared to an antidepressant alone
To evaluate if quetiapine SR in combination with an antidepressant reduces anxiety symptoms in patients with MDD, compared to an antidepressant alone

CONTACTS AND LOCATIONS:
Overall Officials: Seroquel Medical Science Director, MD, Study Director — AstraZeneca
Locations (56):
- United States (56):
  - Research Site, Phoenix, Arizona
  - Research Site, El Centro, California
  - Research Site, Irvine, California
  - Research Site, Oceanside, California
  - Research Site, San Diego, California
  - Research Site, Pueblo, Colorado
  - Research Site, Coral Springs, Florida
  - Research Site, DeLand, Florida
  - Research Site, Gainsville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Roswell, Georgia
  - Research Site, Hoffman Estates, Illinois
  - Research Site, Naperville, Illinois
  - Research Site, Oak Brook, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Lafayette, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Prairie Village, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Shreveport, Louisiana
  - Research SIte, Glen Burnie, Maryland
  - Research Site, Braintree, Massachusetts
  - Research Site, Springfield, Massachusetts
  - Research Site, Clinton Township, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Royal Oak, Michigan
  - Research Site, Saint Charles, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Cherry Hill, New Jersey
  - Research Site, Clementon, New Jersey
  - Research Site, Cedarhurst, New York
  - Research Site, New York, New York
  - Research Site, Olean, New York
  - Research Site, Rochester, New York
  - Research Site, Staten Island, New York
  - Research Site, Beechwood, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Lincoln, Rhode Island
  - Research Site, Columbia, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Friendswood, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research SIte, Wichita Falls, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Arlington, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Bellevue, Washington

REFERENCES:
- [Derived] McIntyre RS, Gorwood P, Thase ME, Liss C, Desai D, Chen J, Bauer M. Early Symptom Improvement as a Predictor of Response to Extended Release Quetiapine in Major Depressive Disorder. J Clin Psychopharmacol. 2015 Dec;35(6):706-10. doi: 10.1097/JCP.0000000000000416. PMID 26474010
- [Derived] Weisler R, Montgomery SA, Earley WR, Szamosi J, Eriksson H. Extended release quetiapine fumarate in patients with major depressive disorder: suicidality data from acute and maintenance studies. J Clin Psychiatry. 2014 May;75(5):520-7. doi: 10.4088/JCP.13m08624. PMID 24816198
- [Derived] Weisler R, McIntyre RS, Bauer M. Extended-release quetiapine fumarate in the treatment of patients with major depressive disorder: adjunct therapy. Expert Rev Neurother. 2013 Nov;13(11):1183-200. doi: 10.1586/14737175.2013.846519. PMID 24175721
- [Derived] Bauer M, Demyttenaere K, El-Khalili N, Thase ME, Papakostas GI, Szamosi J, Earley WR, Eriksson H. Pooled analysis of adjunct extended-release quetiapine fumarate in patients with major depressive disorder according to ongoing SSRI or SNRI treatment. Int Clin Psychopharmacol. 2014 Jan;29(1):16-25. doi: 10.1097/YIC.0000000000000011. PMID 24108148
- [Derived] Clayton AH, Locklear JC, Svedsater H, McIntyre RS. Sexual functioning in patients with major depressive disorder in randomized placebo-controlled studies of extended release quetiapine fumarate. CNS Spectr. 2014 Apr;19(2):182-96. doi: 10.1017/S1092852913000631. Epub 2013 Sep 25. PMID 24067192
- [Derived] Bauer M, McIntyre RS, Szamosi J, Eriksson H. Evaluation of adjunct extended-release quetiapine fumarate on sleep disturbance and quality in patients with major depressive disorder and an inadequate response to on-going antidepressant therapy. Int J Neuropsychopharmacol. 2013 Sep;16(8):1755-65. doi: 10.1017/S146114571300031X. Epub 2013 May 14. PMID 23672772
- [Derived] Vieta E, Bauer M, Montgomery S, McIntyre RS, Szamosi J, Earley WR, Eriksson H. Pooled analysis of sustained response rates for extended release quetiapine fumarate as monotherapy or adjunct to antidepressant therapy in patients with major depressive disorder. J Affect Disord. 2013 Sep 5;150(2):639-43. doi: 10.1016/j.jad.2013.01.052. Epub 2013 Mar 14. PMID 23497790
- [Derived] El-Khalili N, Joyce M, Atkinson S, Buynak RJ, Datto C, Lindgren P, Eriksson H. Extended-release quetiapine fumarate (quetiapine XR) as adjunctive therapy in major depressive disorder (MDD) in patients with an inadequate response to ongoing antidepressant treatment: a multicentre, randomized, double-blind, placebo-controlled study. Int J Neuropsychopharmacol. 2010 Aug;13(7):917-32. doi: 10.1017/S1461145710000015. Epub 2010 Feb 23. PMID 20175941